CLINICAL TRIAL: NCT01064271
Title: A Relative Bioavailability Study of Two Risperidone 1 mg Tablet Formulations Under Fed Conditions
Brief Title: Risperidone Tablets, 1 mg Bioequivalence Study of Dr.Reddy's Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Senior Director - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10640602
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone (Experimental): Risperidone Tablets 1 mg of Dr Reddys Laboratories Limited
  Interventions: Drug: Risperidone
- Risperdal® (Active Comparator): Risperdal® Tablets, 1 mg of Janssen Pharmaceutica Products, L.P
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — Risperidone Tablets 1 mg
  Other Names: Risperdal® Tablets, 1 mg

SUMMARY:
A Single-dose, Randomized, two-Period, Cross over Study

DETAILED DESCRIPTION:
Randomized, single-dose, two-treatment, two-way, crossover study was conducted to compare the relative bioavailability of two risperidone 1 mg tablet formulations under Fed conditions.

The test formulation was Dr. Reddy's Laboratories Limited's 1 mg Risperidone tablet, and the reference formulation was Risperdal® (risperidone) 1 mg tablet (Janssen Pharmaceutica Products, L.P.).

The study was conducted with 26 healthy adults. In each study period, a single 1 mg dose was administered to the subjects following a standardized high-fat breakfast preceded by an overnight fast of at least 10 hours.

The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. There was a 7-day interval between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 - 55 years of age.
2. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable method of contraception (e.g. condom with spermicide, IUD, hormonal contraceptives) for at least 30 days prior to dosing and during the duration of the study.
3. A body mass index (BMI) of 18-30 kg/m² inclusive as calculated according to Novum Standard Operating Procedures.
4. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
5. Signed and dated informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria:

1. If female, pregnant, lactating or likely to become pregnant during the study.
2. History of allergy or sensitivity to risperidone, or similar drugs, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction.
4. Presence of gastrointestinal disease or history of malabsorption within the last year.
5. History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
6. Presence of a medical condition requiring regular treatment with prescription drugs.
7. Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to initial dosing.
8. Receipt of any drug as part of a research study within 30 days prior to dosing.
9. Drug or alcohol addiction requiring treatment in the past 12 months.
10. Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
11. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
12. Positive test results for drugs of abuse at screening.
13. Positive serum pregnancy test.
14. Subjects who smoke more than 10 cigarettes/day or equivalent tobacco use.
15. Subjects who have been on a special diet during the 28 days prior to dosing
16. Subjects who consume on average more than 3 units of alcohol/day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Bio-equivalence study of Dr Reddys Laboratories Risperidone Tablets 1 mg | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Ann Kennedy, MD, Principal Investigator — Novum Pharmaceutical Research Services, 5900 Penn Avenue, Pittsburgh, PA 15206-3817